CLINICAL TRIAL: NCT07346508
Title: Project SPEED - Streamlined Protocol for Early Engagement and Delivery of HIV Prevention With Long-acting Injectable Cabotegravir: A Nurse-driven Protocol
Acronym: Project SPEED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KC Care Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00089751
Record Dates: First submitted 2025-12-18; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: HIV (Human Immunodeficiency Virus)
Keywords: HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The study is a pragmatic implementation science study. Using a parallel 2-arm, single-blind, hybrid type III, cluster randomized controlled design, we will prospectively evaluate the implementation of a nurse-driven LAI-CAB program at the level of LPHDs in MO, USA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SPEED Intervention Group (Experimental): Participants receiving care at LPHDs randomized to the SPEED intervention:
  Interventions: Other: nurse-driven protocol for delivering Long-acting Injectable Cabotegravir (LAI-CAB) for HIV pre-exposure prophylaxis (PrEP)
- Usual PrEP care at Health Departments (No Intervention): Participants receiving care at LPHDs randomized to current practice. The study team will not influence or standardize protocols for care delivery at these LPHDs. Providers will continue to operate based solely on the clinic's usual protocols and provider decisions, without enhancements or additional resources introduced by the study.

INTERVENTIONS:
Other: nurse-driven protocol for delivering Long-acting Injectable Cabotegravir (LAI-CAB) for HIV pre-exposure prophylaxis (PrEP) — Nurse-led PrEP Delivery:
  Nurses assess PrEP eligibility, administer injections, and provide tailored support under established protocols and collaborative practice agreements with medical providers.
  Specialized Training for Nurses:
  Training on sexual health assessments, HIV-risk reduction counseling, PrEP options, injection administration, and identification/reporting of side effects.
  Rapid PrEP Initiation:
  Participants are evaluated for eligibility and receive LAI-CAB within 7 days of enrollment, following CDC guidelines and US prescribing information.
  Comprehensive Care:
  Services include sexual health assessments, rapid HIV testing, STI screening, vaccinations (e.g., HPV, Hepatitis B, MPOX), and HIV/STI risk counseling.
  Medication Procurement and Administration:
  Collaboration with specialty pharmacies for benefits verification, medication procurement, and timely delivery of LAI-CAB to LPHDs for administration.
  Follow-up and Adherence Support:
  Arms: SPEED Intervention Group

SUMMARY:
Project SPEED (Streamlined Protocol for Early Engagement and Delivery of HIV Prevention) is a pragmatic, cluster randomized implementation study evaluating a nurse-driven model for delivering long-acting injectable cabotegravir (LAI-CAB) for HIV pre-exposure prophylaxis (PrEP) within local public health departments (LPHDs) in Missouri. Although LAI-CAB is a highly effective HIV prevention strategy, access remains limited in many rural and resource-constrained settings due to workforce shortages and barriers to specialty care.

In this study, LPHDs are randomized to either implement a structured nurse-led PrEP delivery protocol (SPEED intervention) or continue current standard practices. At intervention sites, trained registered nurses assess PrEP eligibility, provide HIV and sexually transmitted infection testing, administer LAI-CAB injections under standing orders, and support ongoing follow-up as part of routine public health services. Control sites continue their usual workflows without additional training or standardized PrEP delivery processes introduced by the study.

The study uses an effectiveness-implementation hybrid type III design and is guided by established implementation science frameworks to evaluate reach, adoption, implementation, and sustainability of the nurse-driven model. Participants receiving care at participating LPHDs are followed for up to 48 weeks.

Project SPEED aims to generate real-world evidence on whether a nurse-driven approach can expand access to long-acting HIV prevention in public health settings, particularly in rural and underserved communities, and to inform scalable strategies for broader implementation of LAI-CAB PrEP.

DETAILED DESCRIPTION:
Project SPEED (Streamlined Protocol for Early Engagement and Delivery of HIV Prevention) is a pragmatic, hybrid type III effectiveness-implementation study designed to evaluate the adoption, implementation, and sustainability of a nurse-driven model for the delivery of long-acting injectable cabotegravir (LAI-CAB) for HIV pre-exposure prophylaxis (PrEP) within local public health departments (LPHDs) in Missouri. Although LAI-CAB is highly efficacious for HIV prevention, uptake remains limited in the United States, particularly in rural and resource-limited settings where access to licensed prescribers is constrained. This study addresses a critical implementation gap by testing whether trained registered nurses (RNs), operating under protocol-driven supervision and standing orders, can safely and effectively initiate and manage LAI-CAB PrEP services in real-world public health settings.

The study uses a parallel, two-arm, single-blind, cluster randomized controlled design in which LPHDs are the unit of randomization. Participating LPHDs are stratified by geographic and population characteristics (urban, metropolitan, micropolitan, and rural) and randomized in a 1:1 ratio to either the SPEED intervention or current practice. Eight LPHDs are expected to participate, with four assigned to implement the nurse-driven protocol and four continuing usual care. Participants receiving care at these LPHDs are followed for up to 48 weeks.

The SPEED intervention consists of a structured, nurse-led PrEP delivery model that integrates HIV risk assessment, counseling, laboratory testing, vaccination, rapid initiation of PrEP, and ongoing follow-up within routine public health services. RNs at intervention sites are trained to assess PrEP eligibility, conduct HIV and sexually transmitted infection (STI) testing, review laboratory results under standing orders, administer LAI-CAB injections, and provide adherence and risk-reduction counseling. Nurses operate within a collaborative practice framework that includes access to an experienced PrEP provider for consultation when clinically indicated. Rapid PrEP initiation strategies, including short-term oral cabotegravir bridging while insurance approval is pending, are used to minimize delays in starting prevention.

LPHDs assigned to the control arm continue their existing clinical workflows without additional training, protocol changes, or standardized PrEP delivery processes introduced by the study. At these sites, PrEP services, if offered, occur according to local practice, and individuals interested in PrEP may be referred to external providers. Data collection at control sites focuses on documenting current PrEP-related practices and outcomes to allow comparison with intervention sites.

The study is guided by established implementation science frameworks. The Promoting Action on Research Implementation in Health Services (PARIHS) framework informs the implementation strategy, emphasizing the interaction of evidence, context, and facilitation in achieving successful implementation. Evaluation of implementation outcomes is structured using the RE-AIM framework, assessing reach, effectiveness, adoption, implementation, and maintenance at both the participant and organizational levels. Quantitative data from clinical records and surveys are complemented by qualitative interviews with participants and staff to identify barriers, facilitators, and contextual factors influencing implementation.

Project SPEED is designed to generate actionable, real-world evidence on the feasibility, acceptability, and sustainability of nurse-driven LAI-CAB PrEP delivery in public health settings that serve populations disproportionately affected by HIV. Findings will inform the development of a scalable implementation blueprint to support broader adoption of long-acting PrEP within local public health infrastructures, particularly in rural and underserved communities.

ELIGIBILITY:
Inclusion Criteria:

1. Participant seeking medical care at participating LPHDs for family planning, women's wellness exam, STI evaluation, screening, and treatment, and/or any other medical care services.
2. ≥ 18 years of age. The study's focus is on adults. Adolescents may have unique healthcare access challenges, behavioral factors, and parental consent requirements that could complicate study participation.
3. Has an indication for PrEP per guidelines.
4. Understand the commitment to the study and be willing to participate.

Exclusion Criteria:

1. Recent high-risk HIV exposure in the last month and/or has signs/symptoms consistent with acute HIV infection (such as fever, weight loss, skin rash).
2. Unknown, positive, or indeterminate HIV-1 test result by a test approved by the FDA for the diagnosis of acute HIV-1 infection.
3. Any other contraindications based on the most current US Prescribing information.
4. Currently on LAI-CAB, prior use of oral PrEP is not an exclusion criterion.
5. Patients with mental health conditions that are severe enough to interfere with understanding of PrEP requirements (adherence, follow-up visits). The exclusion does not prevent these patients from receiving standard care at the LPHDs; it only excludes them from research-related activities.
6. Inability to provide informed consent, such as due to cognitive or language barriers that prevent understanding of the study requirements.
7. Institutionalized in prison, jail, or healthcare facility. Participants who are institutionalized are excluded because their autonomy may be restricted. Institutional settings also pose logistical challenges for ensuring follow-up and consistent participation in study-related activities.
8. Patients who do not have a confirmed means of contact. Participants must have a reliable means of contact (e.g., phone) to receive laboratory test results, follow-up reminders, and study-related communications.
9. Planning to move out of the area for the follow-up duration of the study. Justification: participants planning to move out of the area cannot reliably complete the study's follow-up visits, which could result in incomplete data.
10. Concurrent participation in another clinical trial. Participants enrolled in other clinical trials may face conflicting protocols, treatment regimens, or follow-up schedules, which could confound study results, introducing biases or safety concerns.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Reach: Did the target population participate in the intervention? | 2 years
  Compare the proportion of participants who started on LAI-CAB during the study period per study arm.

SECONDARY OUTCOMES:
Effectiveness: How effective was the intervention in reducing HIV-1 incidence rates? | 2 years
  HIV-1 incidence rates per 100 person-years adjusted for sexual risk behavior in intervention group versus standard care

OTHER OUTCOMES:
▪ Adoption: How much did the target population accept the intervention and use it? | 18 months
  o To evaluate the acceptability of clinical care associated with the SPEED intervention as reported by participants using the Acceptability Intervention Measure (AIM) at Week 24 and to assess changes in AIM from Week 24 to end of study

IPD SHARING:
Plan to Share IPD: No